CLINICAL TRIAL: NCT03174327
Title: Evaluation of Hepatic Rigidity by Ultrasonic Impulse Elastography in Liver Transplant Patients (SUPERSONIC)
Brief Title: Evaluation of Hepatic Rigidity by Ultrasonic Impulse Elastography in Liver Transplant Patients
Acronym: SUPERSONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC17_9881_SUPERSONIC
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hepatic Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic Transplantation (Other)
  Interventions: Diagnostic Test: Hepatic Transplantation

INTERVENTIONS:
Diagnostic Test: Hepatic Transplantation — Systematic long-term monitoring of liver transplant patients includes an annual consultation and more comprehensive follow-up at one year, 5 years and 10 years of transplantation during which patients are hospitalized in day hospital hepatology and have a clinical examination Complete, biological assessment, Fibroscan® graft elastography measurement, hepatic Doppler ultrasound and liver biopsy. Measurement of liver stiffness by SuperSonic® will be added during ultrasound.
  Other Names: Supersonic® , Fibroscan andHepatic Puncture-Biopsy

SUMMARY:
Interventional study with minimal risks and constraints, prospective, mono-centric.

DETAILED DESCRIPTION:
Ultrasonic impulse elastography is a technique for studying non-invasive tissue rigidity. In particular, it is used in hepatology to assess the degree of fibrosis in a simple manner, by eliminating, in a number of cases, liver biopsy. The investigation of fibrosis is an essential element in the follow-up of patients with hepatic transplant since it is the indirect sign of a post-transplant complication or a recurrence of the initial disease.

Several elastography devices are available on the market, using different technologies to measure the rigidity of tissues. Studies have shown that the first hepatic elastography devices, Fibroscan® and Acoustic Radiation Force Impulse (ARFI) can detect significant fibrosis on hepatic grafts accurately and reproducibly. However, there are several factors related to patients or to the elastography apparatus itself, limiting its use by making the collection of measurements impossible or by giving outliers. In addition, first-generation devices (Fibroscan®) are not coupled to a conventional ultrasound system and are dedicated to the measurement of hepatic rigidity, so patients must undergo systematic ultrasound as part of graft follow-up .

Supersonic® (SuperSonic Imagine, Aix-en-Provence, France) is part of the latest generation of elastography devices and is based on ultrafast shearwave elastography (SWE) technology. This device is a conventional ultrasound system for routine ultrasound scanning with an integrated module for measuring tissue stiffness, and has the advantage of establishing real-time mappings of tissue rigidity over a large area. Several studies have shown that the measurements were reliable and reproducible, especially in the assessment of liver stiffness. In the literature, only one study addressed the measurement of hepatic rigidity with the Supersonic® ultrasound system in liver transplant patients and was designed to diagnose viral hepatitis recurrence or acute cellular rejection. In the secondary results, the authors found a significantly higher hepatic rigidity of healthy hepatic grafts compared to healthy native livers.

It is proposed to add to the ultrasound of systematic follow-up of the hepatic grafts carried out in clinical routine an elastographic measurement in order to assess the hepatic rigidity in these patients in a non-invasive way.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and over ;
* Hepatic transplant patient attending a day hospital of hepatology as part of the systematic follow-up of liver transplantation at 1 year, 5 years or 10 years in order to benefit from a clinical examination, biological evaluation, hepatic ultrasound, Fibroscan and Hepatic Puncture-Biopsy ;
* Patient in a position to receive information about the protocol ;
* Patient having given his / her written consent.

Exclusion Criteria:

* Coagulation disorder (platelets <60,000, Prothrombin Ratio <50%, partial thromboplastin time > 1.5 times the control unless explained by insufficient factor XII deficiency or anti-phospholipid antibodies);
* Ascites;
* Platelet antiaggregation taken the previous week biopsy, patient under anticoagulants;
* Persons of full age who are subject to legal protection (safeguard of justice, guardianship, guardianship), persons deprived of their liberty;
* Patient not affiliated to social security;
* Pregnant or nursing women;
* Simultaneous participation in another research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Hepatic graft stiffness in kPa without complication | Baseline
  Average of the three measures taken consecutively

SECONDARY OUTCOMES:
Hepatic graft stiffness in kPa with complication | Baseline
  Average of the three measures taken consecutively
The performance indicator | Baseline
  Evaluation of the diagnostic performance of Supersonic® and Fibroscan versus Hepatic Puncture-Biopsy (sensitivity, specificity, reproducibility).
The value of the hepatic steatosis of the grafts in the form of a ratio | Baseline
  The value of the hepatic steatosis of the grafts in the form of a ratio between the hepatic brightness and the renal brightness.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Paisant, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dubois M, Ronot M, Houssel-Debry P, Brun V, Rayar M, Auger M, Beuzit L, Turlin B, Aube C, Paisant A. Performance of B-mode ratio and 2D shear wave elastography for the detection and quantification of hepatic steatosis and fibrosis after liver transplantation. Eur J Gastroenterol Hepatol. 2020 Feb;32(2):222-230. doi: 10.1097/MEG.0000000000001500. PMID 31464783